CLINICAL TRIAL: NCT02975037
Title: Evaluation and Validation of Metabolic Markers for the Prediction of Drug-drug Interaction of Various CYP3A4 Substrates and Inhibitors in Healthy Male Subjects
Brief Title: Evaluation of Metabolic Markers for the Prediction of DDI of Various CYP3A Substrates and Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joo-Youn Cho, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CYP3A_DDI
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Healthy
MeSH Terms: interventions — Sildenafil Citrate; Clarithromycin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sildenafil+clarithromycin (Experimental): Sildenafil 25 mg PO (single dose); Clarithromycin 250 mg PO (3 doses); Sildenafil 25 mg PO + Clarithromycin 250 mg PO (single dose)
  Interventions: Drug: Sildenafil; Drug: Clarithromycin
- sildenafil+itraconazole (Experimental): Sildenafil 25 mg PO (single dose); Itraconazole 100 mg PO (3 doses); Sildenafil 25 mg PO + Itraconazole 100 mg PO (single dose)
  Interventions: Drug: Sildenafil; Drug: Itraconazole

INTERVENTIONS:
Drug: Sildenafil — sildenafil 25 mg PO
  Other Names: VIAGRA TAB, Pfizer Pharmaceuticals Korea Limited, Korea
Drug: Clarithromycin — clarithromycin 250 mg PO
  Other Names: CLARI TAB, Hanmi Pharm.Co.,Ltd., Korea
  Arms: sildenafil+clarithromycin
Drug: Itraconazole — itraconazole 100 mg PO
  Other Names: ITRA TAB, Hanmi Pharm.Co.,Ltd., Korea
  Arms: sildenafil+itraconazole

SUMMARY:
Evaluation and validation of metabolic markers for the prediction of drug-drug interaction of various CYP3A4 substrates (sildenafil) and inhibitors (erythromycin/itraconazole) in healthy male subjects

DETAILED DESCRIPTION:
Subjects suitable for this study will be admitted to the Clinical Trials Center, Seoul National University Hospital on the day before dosing, and they will be overnight-fasted from 9P of Day -1. Urine collection is scheduled from 12 hours before sildenafil administration to 12 hours after administration. Subjects will be administered sildenafil (oral) around at 9A of Day 1. Subjects will perform scheduled procedures including clinical laboratory tests, electrocardiograms and blood samplings for pharmacokinetic, pharmacometabolomic and mRNA assessment.

Subjects will be administered either erythromycin or itraconazole (oral) around at 9A on Day 3 and 9A/9P on Day 4. Urine collection is scheduled from 0 hour to 12 hours after Day 3 erythromycin or itraconazole administration. Subjects will perform scheduled procedures including clinical laboratory tests, electrocardiograms and blood samplings for pharmacokinetic, pharmacometabolomic and mRNA assessment.

On Day 5, sildenafil will be administered with erythromycin or itraconazole around at 9A. Urine collection is scheduled from 12 hours before Day 5 drug administration to 12 hours after administration. Subjects will perform scheduled procedures. After subjects perform scheduled procedure, the study will be discharged (around 9A of Day 6).

Study participation was terminated on post-study visit (Day 12-14).

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 19 to 50 years of age, inclusive
* Weight: within 17-28 of Body Mass Index (BMI)
* Subject who are reliable and willing to make themselves available during the study period.
* Subject who are willing to follow the study protocol, and give their written informed consent voluntarily.

Exclusion Criteria:

* History of hypersensitive reaction to medication (midazolam, itraconazole, rifampicin)
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease
* History or evidence of drug abuse
* Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (if used medication is considered acceptable by investigator, patients can be included)
* Participation in clinical trials of any drug within 3 months prior to the participation of the study
* Judged to be inappropriate for the study by the investigator

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-03-04 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Quantification of endogenous metabolites (plasma) | day 1 0h, day 3 0h, day 5 0h
  Metabolomic profiles to predict CYP3A activity
Quantification of endogenous metabolites (urine) | day -1 12h~day 1 0h, day 1 0h~12h, day 3 0h~12h, day 4 12h~ day 5 0h, day 5 0h~12h
  Metabolomic profiles to predict CYP3A activity

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | day 1 0h (pre-dose), 10, 20, 30, 45 min, 1, 2, 3, 4, 6, 8, 12, 24h; day 3 0h (pre-dose), 10, 20, 30, 45 min, 1, 2, 3, 4, 6, 8, 12, 24h; day 5 0h (pre-dose), 10, 20, 30, 45 min, 1, 2, 3, 4, 6, 8, 12, 24h
  Pharmacokinetics of CYP3A substrate and inhibitors
Area under the plasma concentration versus time curve (AUC) | day 1 0h (pre-dose), 10, 20, 30, 45 min, 1, 2, 3, 4, 6, 8, 12, 24h; day 3 0h (pre-dose), 10, 20, 30, 45 min, 1, 2, 3, 4, 6, 8, 12, 24h; day 5 0h (pre-dose), 10, 20, 30, 45 min, 1, 2, 3, 4, 6, 8, 12, 24h
  Pharmacokinetics of CYP3A substrate and inhibitors

OTHER OUTCOMES:
Quantification of mRNA (whole blood) | day -1 12h, day 1 0, 12h, day 3 0, 12h, day 4 12h, day 5 0, 12h
  Quantification of mRNA for CYP3A activity

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Youn Cho, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No